CLINICAL TRIAL: NCT01899859
Title: A Multi-Center, Partially Blinded, Maximum Tolerated Multiple Dose Escalation, Phase 1 Clinical Trial to Evaluate the Safety of GR-MD-02 in Subjects With Non-Alcoholic Steatohepatitis (NASH)With Advanced Hepatic Fibrosis
Brief Title: Phase 1 Study to Evaluate Safety of GR-MD-02 in Subjects With Non-Alcoholic Steatohepatitis (NASH) and Advanced Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galectin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GT-020
Record Dates: First submitted 2013-07-09; First posted 2013-07-16 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2014-06

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH)
Keywords: Non-Alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — belapectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Active Comparator): Patient receives dose of GR-MD-02 or placebo
  Interventions: Drug: GR-MD-02; Drug: Placebo
- Cohort 2 (Active Comparator): Patient receives dose of GR-MD-02 or Placebo
  Interventions: Drug: GR-MD-02; Drug: Placebo
- Cohort 3 (Active Comparator): Patient receives dose of GR-MD-02 or placebo
  Interventions: Drug: GR-MD-02; Drug: Placebo

INTERVENTIONS:
Drug: GR-MD-02 — GR-MD-02; galactoarabino-rhamnogalaturonate
  Other Names: galactoarabino-rhamnogalaturonate
Drug: Placebo — GR-MD-02 Placebo

SUMMARY:
The primary objective of this study is to characterize the safety, tolerability and dose-limiting toxicities (DLTs) for GR-MD-02 when administered intravenously to subjects with biopsy-proven NASH with advanced liver fibrosis.

DETAILED DESCRIPTION:
This study is a dose ranging study to assess in sequential fashion, the safety, tolerability, and dose limiting toxicities (DLTs) of GR-MD-02, in subjects with biopsy-proven NASH with advanced fibrosis. This is a dose escalation design comprised of 3 sequential cohorts to evaluate the safety of GR MD 02 when administered as a single IV infusion followed by 3 additional weekly infusions starting 28 days after the first dose. Each cohort will consist of 8 subjects, 6 randomized to receive active drug and 2 randomized to receive placebo.Based on data safety monitoring board (DSMB) and FDA review, 2 additional cohorts may be implemented, consisting of 8 subjects.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria will be considered for admission to the study:

1. Institutional Review Board (IRB approved written Informed Consent and privacy language as per national regulation (eg, Health Insurance Portability and Accountability Act [HIPAA] Authorization for US sites) must be obtained from the subject or legally authorized representative prior to any study related procedures, including screening evaluations and tests.
2. Subject is ≥ 18 years of age and < 75 years old at the time of consent.
3. Subject has had a percutaneous liver biopsy within 12 months from Screening that shows a definitive diagnosis of NASH with advanced (Brunt stage 3) hepatic fibrosis.
4. Sexually active males and females of childbearing potential must agree to use adequate contraception (condoms, intra-uterine contraceptive device, implants, injectables, sexual abstinence or vasectomized partner) throughout their participation in this study and for 30 days after the last dose of study drug. Women of childbearing potential must have a negative urine pregnancy test within 7 days prior to the first dose. Post-menopausal women must have been amenorrheic for at least 12 months to be considered of non-child-bearing potential.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Subject is a pregnant or lactating female.
2. Subject with current, significant alcohol consumption or a history of significant alcohol consumption for a period of more than 3 consecutive months any time within 1 year prior to screening. Significant alcohol consumption is defined as more than 20 gram per day in females and more than 30 grams per day in males, on average (a standard drink in the US is considered to be 14 grams of alcohol).
3. Subject is unable to reliably quantify alcohol consumption based upon local study physician judgment.
4. Subject uses drugs historically associated with nonalcoholic fatty liver disease (NAFLD) (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, and other known hepatotoxins) for more than 2 weeks in the year prior to Screening.
5. Subject requires use of drugs with a narrow therapeutic window metabolized by CYP3A4 such as fast acting opioids (alfentanil and fentanyl), immunosuppressive drugs (cyclosporine, sirolimus, and tacrolimus), some cardiovascular agents (ergotamine, quinidine and dihydroergotamine), and select psychotropic agents (pimozide).
6. Subject has prior or has planned (during the study period) bariatric surgery (eg, gastroplasty, Roux-en-Y gastric bypass).
7. Subject has concurrent infection including diagnoses of fever of unknown origin and evidence of possible central line sepsis (subjects must be afebrile at the start of therapy).
8. Subject with a platelet count below 100,000/mm3 at Screening.
9. Subject with clinical evidence of hepatic decompensation as defined by the presence of any of the following abnormalities at Screening:

   1. Serum albumin less than 3.5 grams/deciliter (g/dL).
   2. An INR greater than 1.1.
   3. Direct bilirubin greater than 1.3 milligrams per deciliter (mg/dL).
10. Subject has a history of bleeding esophageal varices, ascites or hepatic encephalopathy
11. Subject has a history of hepatitis C. Patients found on screening to have hepatitis C antibody, even if PCR negative for HCV RNA, are excluded from this study.
12. Subject has evidence of other forms of chronic liver disease:

    1. Hepatitis B as defined by presence of hepatitis B surface antigen.
    2. Evidence of ongoing autoimmune liver disease as defined by compatible liver histology.
    3. Primary biliary cirrhosis as defined by the presence of at least 2 of these criteria (i) Biochemical evidence of cholestasis based mainly on alkaline phosphatase elevation (ii) Presence of anti-mitochondrial antibody (iii) Histologic evidence of nonsuppurative destructive cholangitis and destruction of interlobular bile ducts.
    4. Primary sclerosing cholangitis.
    5. Wilson's disease as defined by ceruloplasmin below the limits of normal and compatible liver histology.
    6. Alpha-1-antitrypsin deficiency as defined by diagnostic features in liver histology (confirmed by alpha-1 antitrypsin level less than normal; exclusion at the discretion of the study physician).
    7. History of hemochromatosis or iron overload as defined by presence of 3+ or 4+ stainable iron on liver biopsy.
    8. Drug-induced liver disease as defined on the basis of typical exposure and history.
    9. Known bile duct obstruction.
    10. Suspected or proven liver cancer.
    11. Any other type of liver disease other than NASH.
13. Subject with serum ALT greater than 300 units per liter (U/L) at Screening.
14. Subject with serum creatinine of 1.5 mg/dL or greater at Screening.
15. Subject using of any prescription or over-the-counter medication or herbal remedy that are believed to improve or treat NASH or liver disease or obesity during the period beginning 30 days prior to randomization. Subjects who are using Vitamin E or omega-3 fatty acids may continue their use.
16. Subject had major surgery within 8 weeks prior to Day 0, significant traumatic injury, or anticipation of need for major surgical procedure during the course of the study.
17. Subject with a history of biliary diversion.
18. Subject with known positivity for Human Immunodeficiency Virus infection.
19. Subject with an active, serious medical disease with likely life expectancy of less than 5 years.
20. Subject with active substance abuse, including inhaled or injection drugs, in the year prior to Screening.
21. Subject who has clinically significant and uncontrolled cardiovascular disease (eg, uncontrolled hypertension, myocardial infarction, unstable angina), New York Heart Association Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or Grade II or greater peripheral vascular disease within 12 months prior to Day 0.
22. Subject has participated in an investigational new drug (IND) trial in the 30 days before randomization.
23. Subject has a clinically significant medical or psychiatric condition considered a high risk for participation in an investigational study.
24. Subject has any other condition which, in the opinion of the Investigator, would impede compliance or hinder completion of the study.
25. Subject has been previously exposed to GR MD 02.
26. Subject with known allergies to the study drug or any of its excipients.
27. Subject with malignant disease (other than basal and squamous cell carcinoma of the skin and in situ carcinoma of the cervix) with at least 5 years of follow-up showing no recurrence.
28. Subject has an abnormal chest x-ray indicative of acute or chronic lung disease on screening examination.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Primary objective is to characterize safety for GR-MD-02 administered intravenously to subjects w/ biopsy-proven NASH w/ advanced liver fibrosis. Specifically assessed by number of subjects experiencing TEAEs. | Baseline; Week 1-7 (End of Study); Week 9; Week 11 (Follow-up)
  The primary objective of this study is to characterize the safety, which includes the tolerability and dose-limiting toxicity (DLT), for GR-MD-02 when administered intravenously to subjects with biopsy-proven NASH with advanced liver fibrosis. Specifically, this measure will be assessed by number of subjects experiencing treatment emergent adverse events indicative of DLT.

SECONDARY OUTCOMES:
A secondary objective is to characterize the first-dose PK profile of GR-MD-02. The PK profile is assessed by the AUC (area under the plasma concentration versus time curve) and Cmax (peak plasma concentration) of GR-MD-02. | Baseline; Week 1-4
  A secondary objective for the study is to characterize the first-dose PK profile of GR-MD-02 administered as an IV infusion. Specifically, the PK profile is assessed by the AUC (area under the plasma concentration versus time curve) and Cmax (peak plasma concentration) of GR-MD-02.
A secondary objective for the study is to characterize the PK profile and serum level accumulation of GR-MD-02 following administration of 3 subsequent weekly doses given by IV infusion beginning 28 days after the first dose. | Baseline; Week 5-7 (End of Study)
  A secondary objective for the study is to characterize the PK profile and serum level accumulation of GR-MD-02 following administration of 3 subsequent weekly doses given by IV infusion beginning 28 days after the first dose.
A secondary objective is to evaluate change in serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), ratio of AST:ALT, alkaline phosphatase, and gamma glutamyl transpeptidase (GGTP); change in AST/platelet ratio index. | Baseline; Week 7 (End of Study)
  A secondary objective for this study is to evaluate change in serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), ratio of AST:ALT, alkaline phosphatase, and gamma glutamyl transpeptidase (GGTP) levels; and change in AST/platelet ratio index.
A secondary objective for this study is to evaluate changes in exploratory pharmacodynamic biomarkers in serum | Baseline; Week 7 (End of Study)
  A secondary objective for this study is to evaluate levels of exploratory pharmacodynamic biomarkers in serum including galectin-3, inflammatory, cell-death, and fibrosis markers.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Harrison, MD, Principal Investigator — Brooke Army Medical Center; Naga Chalasani, MD, Principal Investigator — Indiana University School of Medicine; Ram Subramanian, MD, Principal Investigator — Emory University Hospital (Transplant Center Clinical Research); Thomas Schiano, MD, Principal Investigator — The Mount Sinai Medical Center (Division of Liver Diseases); Brent A Tetri, MD, Principal Investigator — St. Louis University School of Medicine; Mohammad S Siddiqui, MD, Principal Investigator — Virginia Commonwealth University Medical Center
Locations (1):
- Brooke Army Medical Ctr., San Antonio, Texas, United States

REFERENCES:
- [Derived] Machado MV, Diehl AM. Liver renewal: detecting misrepair and optimizing regeneration. Mayo Clin Proc. 2014 Jan;89(1):120-30. doi: 10.1016/j.mayocp.2013.10.009. PMID 24388030